CLINICAL TRIAL: NCT06676800
Title: Observation Study on the Efficacy of Yiqi Gubiao Pill in the Treatment of Chronic Obstructive Pulmonary Disease Secondary to Active Pulmonary Tuberculosis: A Double-Blind Randomized Controlled Trial Protocol
Brief Title: Observation Study on the Efficacy of Yiqi Gubiao Pill in the Treatment of Chronic Obstructive Pulmonary Disease Secondary to Active Pulmonary Tuberculosis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fourth Affiliated Hospital of Xinjiang Medical University (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jin Dai, Attending Physician, Fourth Affiliated Hospital of Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021D01C215
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis-related Obstructive Pulmonary Disease
Keywords: Pulmonary tuberculosis; Yiqi Gubiao Pills; Chronic Obstructive Pulmonary Disease; Randomized double-blind placebo-controlled trial
MeSH Terms: conditions — Tuberculosis, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yiqi Gubiao pill (Experimental)
  Interventions: Drug: Yiqi Gubiao pill
- Yiqi Gubiao Pill placebo (Placebo Comparator)
  Interventions: Drug: Yiqi Gubiao Pill placebo

INTERVENTIONS:
Drug: Yiqi Gubiao pill — Take 10 pills orally each time, three times a day, after meals, for a continuous period of 12 weeks. Receiving basic treatment: standardized quadruple anti-tuberculosis therapy is administered, with Rifampicin, Isoniazid, Ethambutol, and Pyrazinamide used for the first 2 months, followed by Rifampicin and Isoniazid for the next 4 months.
  Arms: Yiqi Gubiao pill
Drug: Yiqi Gubiao Pill placebo — The placebo's appearance and content color are similar to that of Yiqi Gubiao Pill, with the main ingredients being starch and caramel. Take 10 pills orally each time, three times a day, after meals, for a continuous period of 12 weeks. Receiving basic treatment: standardized quadruple anti-tuberculosis therapy is administered, with Rifampicin, Isoniazid, Ethambutol, and Pyrazinamide used for the first 2 months, followed by Rifampicin and Isoniazid for the next 4 months.
  Arms: Yiqi Gubiao Pill placebo

SUMMARY:
Tuberculosis-related obstructive pulmonary disease (TOPD), as a high-burden disease in most countries, poses difficulties in the diagnosis and treatment of the disease when coexisting, and increases the risk of death for patients. Preliminary studies have shown that Yiqi Gubiao Wan has significant effects in relieving cough, alleviating asthma, expectorating phlegm, and delaying airway obstruction. The purpose of this study is to verify the therapeutic effect of Yiqi Gubiao pill on patients with TOPD through rigorous methodological design and to evaluate its safety. We will conduct a prospective, double-blind, randomized controlled trial. First, participants will be randomly assigned 1:1 to the Yiqi Gubiao pill treatment group and the Yiqi Gubiao pill placebo control group. This will be followed by a 12-week treatment. During the treatment period, we will measure and record the patients' lung function and quality of life. We will also score the patients' TCM symptoms. Finally, the safety of the medication will be assessed.

ELIGIBILITY:
Inclusion Criteria:

-

Patients who meet the following criteria will be included:

1. Age 40-75 years old;
2. Meet the Western medical diagnostic criteria and typing standards for active PTB;
3. Patients who have not taken steroids, anti-tuberculosis drugs, or other immunosuppressants and have not undergone desensitization treatment within one month.
4. Have understood the treatment methods and voluntarily signed the informed consent form.

Exclusion Criteria:

-

Patients who meet any of the following criteria will be excluded:

1. Patients with pneumothorax, pleural effusion, lung cancer and other serious lung diseases;
2. Patients with severe cardiovascular and cerebrovascular, hepatorenal and hematopoietic diseases;
3. mentally ill;
4. Patients with tumors;
5. Congenital or acquired immunodeficiency.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity | up to 4 weeks
  Forced Vital Capacity (FVC) refers to the volume of air exhaled as quickly and forcefully as possible after taking the maximum inhalation.
the percentage of FVC predicted | up to 4 weeks
  The volume of air exhaled rapidly within one second after inhaling to the total lung capacity. Normal values are 70-85%, mild is less than 80% of the predicted value; moderate is less than 70% of the predicted value; moderately severe is less than 60% of the predicted value; severe is less than 50% of the predicted value.
the ratio of FEV1 to FVC | up to 4 weeks
  The ratio of FEV1 to FVC should be above 70%. If the ratio is below 70%, it may indicate the presence of chronic obstructive pulmonary disease (COPD).
COPD Assessment Test (CAT) score | up to 4 weeks
  The CAT score questionnaire is primarily used to assess the health status and impact on daily life of patients with chronic obstructive pulmonary disease (COPD). It quantifies the degree of health impairment in COPD patients by asking questions related to symptoms, activity ability, mental state, and social impact based on the patients' self-reports. The total score of the CAT questionnaire ranges from 0 to 40, with higher scores indicating poorer health status and lower quality of life for the patients.
modified Medical Research Council (mMRC) score | up to 4 weeks
  The mMRC is only used for the assessment of dyspnea and is often applied in conjunction with the CAT score. An mMRC score of 2 or above is the threshold for distinguishing "mild dyspnea" from "severe dyspnea."
Baseline Dyspnea Index (BDI) score | up to 4 weeks
  It measures activity-related dyspnea from three dimensions: degree of functional impairment, amount of activity, and effort required to complete activities. Each dimension is graded on a 5-level scale, with scores ranging from 0 to 4, indicating increasing severity. The total score ranges from 0 to 12.
Transition Dyspnea Index (TDI) score | up to 4 weeks
  The TDI should be used in conjunction with the BDI to measure the extent of change in prognostic functional impairment, activity level, and effort required to complete activities. The TDI scores each dimension on a scale from significantly worse (-3) to significantly better (+3), with a total score ranging from -9 to +9.

SECONDARY OUTCOMES:
Traditional Chinese Medicine (TCM) symptom score | up to 4 weeks
  The main symptoms and secondary symptoms are graded from mild to severe into 4 levels. The main symptoms are scored 0, 2, 4, 6 points respectively, and the secondary symptoms are scored 0, 1, 2, 3 points respectively. The tongue and pulse are not scored. The sum of the scores for all symptoms is the total TCM symptom score.
alanine aminotransferase | up to 4 weeks
  The reference range is 0-40 U/L.
aspartate aminotransferase | up to 4 weeks
  The reference range is 0-40 U/L.
urea nitrogen | up to 4 weeks
  Reference range value 3.2-7.1 mmol/L
serum creatinine | up to 4 weeks
  Reference range value: Males 53-106 μmol/L, Females 44-97 μmol/L
uric acid | up to 4 weeks
  Normal serum uric acid values: for adult males, 149-416 μmol/L; for adult females, 89-357 μmol/L.

REFERENCES:
- [Background] Bagcchi S. WHO's Global Tuberculosis Report 2022. Lancet Microbe. 2023 Jan;4(1):e20. doi: 10.1016/S2666-5247(22)00359-7. Epub 2022 Dec 12. No abstract available. PMID 36521512
- [Derived] Dai J, Zhang Y, Su J, Yuan G, Li F, Zhou Z, Aziza, Ye C, Seyiti A, Pida M, Zhang J. Yiqi Gubiao Pill for tuberculosis-associated obstructive pulmonary disease: protocol for a double-blind randomized controlled trial. Front Pharmacol. 2025 Oct 8;16:1610889. doi: 10.3389/fphar.2025.1610889. eCollection 2025. PMID 41132532